CLINICAL TRIAL: NCT02592551
Title: Window Of Opportunity Phase II Study Of MEDI4736 Or MEDI4736 + Tremelimumab In Surgically Resectable Malignant Pleural Mesothelioma
Brief Title: MEDI4736 Or MEDI4736 + Tremelimumab In Surgically Resectable Malignant Pleural Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Bryan Burt, MD, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H-36952
Record Dates: First submitted 2015-10-19; First posted 2015-10-30 (Estimated); Results first posted 2022-01-13 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Mesothelioma
MeSH Terms: conditions — Mesothelioma | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MEDI4736 (Experimental): 8 patients will receive an infusion of MEDI4736 (15 mg/kg intravenously, once), one to six weeks prior to surgical resection.
  Interventions: Drug: MEDI4736
- MEDI4736 + Tremelimumab (Active Comparator): 8 patients will receive an infusion of MEDI4736 (1500 mg intravenously, once) + tremelimumab (75mg intravenously, once), one to six weeks prior to surgical resection.
  Interventions: Drug: MEDI4736; Drug: Tremelimumab
- Untreated arm (control) (Placebo Comparator): 4 patients will not receive MEDI4736 or Tremelimumab.
  Interventions: Other: no other name

INTERVENTIONS:
Drug: MEDI4736 — MEDI4736 is formulated at 50 mg/mL in 26 mM histidine/histidine-HCl, 275 mM trehalose dihydrate, 0.02% (w/v) polysorbate 80, pH 6.0.
  Other Names: durvalumab
  Arms: MEDI4736; MEDI4736 + Tremelimumab
Drug: Tremelimumab — Tremelimumab Drug Product is formulated at a nominal concentration of 20 mg/mL in 20 mM histidine/histidine hydrochloride, 222 mM trehalose dihydrate, 0.02% (weight/volume [w/v]) polysorbate 80, 0.27 mM disodium edetate dihydrate (EDTA), pH 5.5.
  Other Names: no other name
  Arms: MEDI4736 + Tremelimumab
Other: no other name — Neither MEDI4736 nor Tremelimumab will be used.
  Arms: Untreated arm (control)

SUMMARY:
The objective of this study is to determine whether MEDI4736 or combination therapy with MEDI4736 + tremelimumab are associated with favorable alterations of the intratumoral immunologic environment in subjects undergoing resectional surgery for Malignant Pleural Mesothelioma MPM.

DETAILED DESCRIPTION:
Subjects with MPM will undergo surgical mediastinal lymph node biopsy (cervical mediastinoscopy) and simultaneous surgical biopsy of the pleural tumor by thoracoscopy, at which time tumor tissue (at least 2 g) and peripheral blood will be collected for the study. These procedures are performed as standard of care in the treatment of these subjects. The subject will be randomized. Three days to three weeks after the biopsy, subjects will be randomly treated with either MEDI-4736 (15 mg/kg once intravenously) or MEDI-4736 (1500 mg once intravenously) plus tremelimumab (75 mg once intravenously) or a control group in a randomized controlled study design. There will be two treatment arms (MEDI4736 only and combination MEDI4736+tremelimumab) and one untreated arm (control). Randomization, stratified by receiving previous chemotherapy or not, will be performed and will help to minimize patient selection biases between three arms. Subjects under 30 kg will be treated with weight-based dosing for both MEDI4736 and Tremelimumab combination therapy. These patients are excluded from fixed based dosing to limit endotoxin exposure from the drug preparations. One to six weeks after the infusion, subjects will undergo resectional surgery, including extrapleural pneumonectomy (EPP) or pleurectomy/decortication (P/D), at which time the tumor will be removed (typically 200-1000 g) and obtained for study. Four patients that do not undergo treatment with MEDI-4736 or tremelimumab will be included as controls. Blood will be obtained after the induction of general anesthesia for both the thoracoscopy procedure and the EPP or P/D resectional procedure, as is routinely done in these procedures. The sixth rib will be obtained at the time of the resection. After the removal of the tumor, standard protocol includes intraoperative heated chemotherapy using a lavage of intracavitary cisplatin in the presence of conserved renal function (Sugarbaker et al., 2013, 2014; Richards et al., 2006).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
2. Age >/= 18 years at time of study entry
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Adequate normal organ and marrow function as defined below:

   Hemoglobin ≥ 9.0 g/dL Absolute neutrophil count (ANC) ≥ 1.5 × 109/L (> 1500 per mm3) Platelet count ≥ 100 × 109/L (>100,000 per mm3) Serum bilirubin ≤ 1.5× institutional upper limit of normal (ULN)AST<3.0 Creatinine clearance >50mL/miN Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 × ULN (≤ 5 × ULN if documented liver metastasis are present); Serum creatinine ≤ 2.0 mg/dL or calculated creatinine clearance ≥ 50 mL/min as determined by the Cockcroft-Gault equation;

   Males:

   Creatinine CL (mL/min) = Weight (kg) × (140 - Age) 72 × serum creatinine (mg/dL)

   Females:

   Creatinine CL (mL/min) = Weight (kg) × (140 - Age) × 0.85 72 × serum creatinine (mg/dL)
5. Female subjects must either be of non-reproductive potential (i.e., post-menopausal by history: ≥60 years old and no menses for >/=1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry.
6. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
7. Surgically resectable MPM with no disease extension beyond the ipsilateral hemithorax
8. Planned resectional surgery for MPM [extrapleural pneumonectomy (EPP) or pleurectomy and decortication (P/D)]
9. Any MPM histology (epithelial, mixed, sarcomatoid)
10. N0 or N1 nodal disease as present on perioperative chest CT and/or PET CT.
11. N2 nodal disease if no progression after 2 cycles of standard chemotherapy. Progression will be considered if additional N1 or N2 disease develop during chemotherapy

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site) or previous enrollment or randomization in the present study
2. Participation in another clinical study with an investigational product during the last 3 months
3. Any previous treatment with a PD1 or PD-L1 inhibitor, including MEDI4736
4. Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) 30 days prior to the first dose of study drug, and 30 days prior to the first dose of study drug for subjects who have received prior TKIs [e.g., erlotinib, gefitinib and crizotinib] and within 6 weeks for nitrosourea or mitomycin C).
5. Current or prior use of immunosuppressive medication within 28 days before the infusion with MEDI4736 or MEDI4736 + tremelimumab and through 90 days post infusion, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid.
6. Any unresolved toxicity (>CTCAE grade 2) from previous anti-cancer therapy.
7. Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1
8. Active or prior documented autoimmune disease within the past 2 years NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
9. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
10. History of primary immunodeficiency
11. History of allogeneic organ transplant
12. History of hypersensitivity to MEDI4736 or any excipient
13. History of hypersensitivity to tremelimumab or the combination of MEDI4736 + tremelimumab
14. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
15. Known history of previous clinical diagnosis of tuberculosis
16. History of leptomeningeal carcinomatosis
17. Receipt of live attenuated vaccination within 30 days prior to study entry or within 6 months of receiving MEDI4736 or MEDI + tremelimumab
18. Receipt of drugs with laxative properties and herbal or natural remedies for constipation within 90 days of receiving MEDI4736 or MEDI + tremelimumab
19. Receipt of sunitinib within 3 months of receiving tremelimumab
20. Female subjects who are pregnant, breastfeeding, or male or female subjects of reproductive potential who are not employing an effective method of birth control
21. Any condition that, in the opinion of the investigator, would interfere with the evaluation of the study treatment or interpretation of subject safety or study results
22. Symptomatic or uncontrolled brain metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation, and/or corticosteroids.
23. Subjects with uncontrolled seizures
24. N3 nodal disease
25. History of interstitial lung disease/pneumonitis
26. No tissue is obtainable at the time of thoracoscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2022-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Burt, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor St Lukes, Houston, Texas, United States

REFERENCES:
- [Derived] Lee HS, Jang HJ, Ramineni M, Wang DY, Ramos D, Choi JM, Splawn T, Espinoza M, Almarez M, Hosey L, Jo E, Hilsenbeck S, Amos CI, Ripley RT, Burt BM. A Phase II Window of Opportunity Study of Neoadjuvant PD-L1 versus PD-L1 plus CTLA-4 Blockade for Patients with Malignant Pleural Mesothelioma. Clin Cancer Res. 2023 Feb 1;29(3):548-559. doi: 10.1158/1078-0432.CCR-22-2566. PMID 36469573

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MEDI4736 | MEDI4736 + Tremelimumab | Untreated Arm (Control)
Started | 9 | 11 | 4
Completed | 8 (One participant completed all study procedures and got the tumor sample for analysis. However, the sample was too small to analyze in the lab and so that it was not evaluable for primary and secondary analysis.) | 8 | 4
Not Completed | 1 | 3 | 0
Not completed — Not evaluable | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all participants enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | MEDI4736 | MEDI4736 + Tremelimumab | Untreated Arm (Control) | Total
Number analyzed (Participants) | 9 | 11 | 4 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (6) | 59 (15) | 58 (12) | 63 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 6
  Male | 7 | 9 | 2 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 3
  Not Hispanic or Latino | 9 | 9 | 3 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 9 | 11 | 1 | 21
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 2
Prior Chemodtherapy [Count of Participants; unit: Participants]
  Yes | 0 | 1 | 2 | 3
  No | 9 | 10 | 2 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Ratio of Intratumoral Cytotoxic T Cells to Regulatory T Cells (CD8/Treg)
Description: Tissue biomarker immune response of CD8 and Treg to before and after MEDI-4736 and Tremelimumab will be obtained using CytoF (time-of-flight mass cytometry) and/or flow cytometry. The ratios of CD8/Treg are calculated by diving CD8 by Treg.
Time Frame: at day 1 after screening and at a surgery within one to six weeks after treatment
Population: The primary objective was the comparison of CD8/Treg before and after treatment with combination MEDI-4736 and Tremelimumab group. Therefore, the analysis population was from one arm (MEDI4736+Tremelimumab).
Measure: Median (Inter-Quartile Range); unit: no unit of ratios with same units(%)
Arm/Group | MEDI4736 + Tremelimumab
Number analyzed (Participants) | 8
no unit of ratios with same units(%) | 8.6 [-1.4 to 29.9]
Statistical Analysis 1: Comparison: MEDI4736 + Tremelimumab; Compare in ratios of intratumoral cytotoxic T cells to regulatory T cells (CD8/Treg) between pre and post of MEDI4736+Tremelimumab; Test type: Other; p = 0.109, Wilcoxon signed rank test; Median Difference (Final Values) = 8.6

2. Secondary Outcome: Change in Percentage of Inducible T-cell Co-stimulator (ICOS) + CD4 T Cells.
Description: Tissue biomarker for the immune response of ICOS+ CD4 T cells to before and after MEDI-4736 and Tremelimumab will be obtained using CytoF (time-of-flight mass cytometry) and/or flow cytometry. The percentages of ICOS+CD4 T cells are calculated by dividing by total cells.
Time Frame: at day 1 after screening and at a surgery within one to six weeks after treatment
Population: The objective was the comparison of percentage of inducible T-cell co-stimulator (ICOS) + CD4 T cells before and after treatment with combination MEDI-4736 and Tremelimumab group. Therefore, the analysis population was from one arm (MEDI4736+Tremelimumab).
Measure: Median (Inter-Quartile Range); unit: percentage of inducible T-cell co-stimul
Arm/Group | MEDI4736 + Tremelimumab
Number analyzed (Participants) | 8
percentage of inducible T-cell co-stimul | -2.1 [-5.2 to 1]
Statistical Analysis 1: Comparison: MEDI4736 + Tremelimumab; Test type: Other — Compare the tissue biomarker for the immune response of ICOS+ CD4 T cells to before and after MEDI-4736 and Tremelimumab; p = 1, Wilcoxon signed rank test

3. Secondary Outcome: Change in Tumor Expression Programmed Death-ligand 1 (PD-L1).
Description: Tumor expression programmed death-ligand 1 (PD-L1) before and after treatment with combination MEDI-4736 and Tremelimumab will be obtained by immunohistochemistry and CytoF. The unit of measure is MMI. MMI (mean metal intensity or mean mass intensity) is a signal intensity in time-of-flight mass cytometry (CyTOF), which is the same as MFI (mean fluorescent intensity) in flow cytometry. Mean metal intensity looks more common in CyTOF to tell it from the unit in mass spectrometry. Its range is from 0 to infinity.
Time Frame: at day 1 after screening and at a surgery within one to six weeks after treatment
Population: The objective was the comparison of tumor expression programmed death-ligand 1 (PD-L1) before and after treatment with combination MEDI-4736 and Tremelimumab group. Therefore, the analysis population was from one arm (MEDI4736+Tremelimumab).
Measure: Median (Inter-Quartile Range); unit: MMI (Mean Mass Intensity)
Arm/Group | MEDI4736 + Tremelimumab
Number analyzed (Participants) | 8
MMI (Mean Mass Intensity) | 0.07 [-0.12 to 0.30]
Statistical Analysis 1: Comparison: MEDI4736 + Tremelimumab; Compare tumor expression programmed death-ligand 1 (PD-L1) before and after treatment with combination MEDI-4736 and Tremelimumab; Test type: Other; p = 0.461, Wilcoxon signed rank test

4. Secondary Outcome: Ratio of Intratumoral Cytotoxic T Cells to Regulatory T Cells (CD8/Treg) in Patients Treated With Combination Therapy (MEDI-4736 and Tremelimumab) and in Patients Treated With MEDI-4736 Alone.
Description: Tissue biomarker immune response of CD8 and Treg after MEDI-4736 and Tremelimumab, and after MEDI4736 alone will be obtained using CytoF (time-of-flight mass cytometry) and/or flow cytometry. The ratios of CD8/Treg are calculated by diving CD8 by Treg.
Time Frame: at a surgery within one to six weeks after treatment
Population: one participant who was assigned to MEDI4736 alone group completed the study procedures but the tumor sample was too small to analyze in the lab.
Measure: Median (Inter-Quartile Range); unit: no unit of ratios with same units(%)
Arm/Group | MEDI4736 | MEDI4736 + Tremelimumab
Number analyzed (Participants) | 7 | 8
no unit of ratios with same units(%) | 8 [3.4 to 9.4] | 9.7 [2 to 20.9]
Statistical Analysis 1: Comparison: MEDI4736 vs MEDI4736 + Tremelimumab; Compare tissue biomarker immune response of CD8 and Treg (ratio of CD8/treg) after MEDI-4736 and Tremelimumab, and after MEDI4736 alone; Test type: Other; p = 0.954, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Ratio of Intratumoral Cytotoxic T Cells to Regulatory T Cells (CD8/Treg) in Patients Treated With Combination Therapy (MEDI-4736 and Tremelimumab) and Untreated Patients.
Description: Tissue biomarker immune response of CD8 and Treg after MEDI-4736 and Tremelimumab, and at day 1 of untread will be obtained using CytoF (time-of-flight mass cytometry) and/or flow cytometry. The ratios of CD8/Treg are calculated by diving CD8 by Treg.
Time Frame: the untreated group(control) : at day 1, MEDI4736 + Tremelimumab: at a surgery within one to six weeks after treatment (MEDI4736+Tremelimumab) group
Measure: Median (Inter-Quartile Range); unit: no unit of ratios with same units(%)
Arm/Group | MEDI4736 + Tremelimumab | Untreated Arm (Control)
Number analyzed (Participants) | 8 | 4
no unit of ratios with same units(%) | 9.7 [2 to 20.9] | 4.03 [2.7 to 12.6]
Statistical Analysis 1: Comparison: MEDI4736 + Tremelimumab vs Untreated Arm (Control); Compare tissue biomarker immune response of CD8 and Treg(ratio of CD8/Treg) after MEDI-4736 and Tremelimumab, and at day 1 of untread control group; Test type: Other; p = 0.799, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Percentage of Inducible T-cell Co-stimulator (ICOS) + CD4 T Cells in Patients Treated With Combination Therapy (MEDI-4736 and Tremelimumab) and in Patients Treated With MEDI-4736 Alone
Description: Tissue biomarker immune response of ICOS+ CD4 T cells after combination therapy (MEDI-4736 and Tremelimumab) and after MEDI4736 alone will be obtained using CytoF (time-of-flight mass cytometry) and/or flow cytometry. The percentages of ICOS+CD4 T cells are calculated by dividing by total cells.
Time Frame: at a surgery within one to six weeks after treatment
Population: Percentages of ICOS(+) CD8 T cells were obtained in only three patients who have enough amount of live single cells in post-treatment tumor samples in MEDI4736 group and in two patient in MEDI4736+Tremelimumab group.
Measure: Median (Inter-Quartile Range); unit: percentage of (ICOS) + CD4 T cells
Arm/Group | MEDI4736 | MEDI4736 + Tremelimumab
Number analyzed (Participants) | 3 | 2
percentage of (ICOS) + CD4 T cells | 1.2 [0.5 to 3.9] | 4.5 [2.5 to 6.5]

7. Secondary Outcome: Percentage of Inducible T-cell Co-stimulator (ICOS) + CD4 T Cells in Patients Treated With Combination Therapy (MEDI-4736 and Tremelimumab) and in Untreated Patients.
Description: Tissue biomarker immune response of ICOS+ CD4 T cells after combination therapy (MEDI-4736 and Tremelimumab) and after untreated patients will be obtained using CytoF (time-of-flight mass cytometry) and/or flow cytometry. The percentages of ICOS+CD4 T cells are calculated by dividing by total cells.
Time Frame: Untreated group (control): at day 1, MEDI-4736 and Tremelimumab group: at a surgery within one to six weeks after treatment
Population: Percentages of ICOS(+) CD8 T cells were obtained in only two patients who have enough amount of live single cells in post-treatment tumor samples in MEDI4736+Tremelimumab group. No patients in the untreated arm had enough cells.
Measure: Median (Inter-Quartile Range); unit: percentage of (ICOS) + CD4 T cells
Arm/Group | MEDI4736 + Tremelimumab | Untreated Arm (Control)
Number analyzed (Participants) | 2 | 0
percentage of (ICOS) + CD4 T cells | 4.5 [2.5 to 6.5] |

8. Secondary Outcome: Tumor Expression Programmed Death-ligand 1 (PD-L1) in Patients Treated With Combination Therapy (MEDI-4736 and Tremelimumab) and in Patients Treated With MEDI-4736 Alone.
Description: Tumor expression programmed death-ligand 1 (PD-L1) after combination therapy (MEDI-4736 and Tremelimumab) and after MEDI-4736 alone will be obtained by immunohistochemistry and CytoF. The unit of measure is MMI. MMI (mean metal intensity or mean mass intensity) is a signal intensity in time-of-flight mass cytometry (CyTOF), which is the same as MFI (mean fluorescent intensity) in flow cytometry. Mean metal intensity looks more common in CyTOF to tell it from the unit in mass spectrometry. Its range is from 0 to infinity.
Time Frame: at a surgery within one to six weeks after treatment
Measure: Median (Inter-Quartile Range); unit: MMI (Mean Mass Intensity)
Arm/Group | MEDI4736 | MEDI4736 + Tremelimumab
Number analyzed (Participants) | 7 | 8
MMI (Mean Mass Intensity) | 0.31 [0.19 to 0.69] | 0.18 [0.12 to 0.59]
Statistical Analysis 1: Comparison: MEDI4736 vs MEDI4736 + Tremelimumab; Compare tumor expression programmed death-ligand 1 (PD-L1) after combination therapy (MEDI-4736 and Tremelimumab) and after MEDI-4736 alone; Test type: Other; p = 0.418, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Tumor Expression Programmed Death-ligand 1 (PD-L1) in Patients Treated With Combination Therapy (MEDI-4736 and Tremelimumab) and in Untreated Patients.
Description: Tumor expression programmed death-ligand 1 (PD-L1) after combination therapy (MEDI-4736 and Tremelimumab) and before and at day 1 of untreate alone will be obtained by immunohistochemistry and CytoF. The unit of measure is MMI. MMI (mean metal intensity or mean mass intensity) is a signal intensity in time-of-flight mass cytometry (CyTOF), which is the same as MFI (mean fluorescent intensity) in flow cytometry. Mean metal intensity looks more common in CyTOF to tell it from the unit in mass spectrometry. Its range is from 0 to infinity.
Time Frame: Untreated arm (control): at day 1 after screening, MEDI4736 + Tremelimumab group: at a surgery within one to six weeks after treatment
Measure: Median (Inter-Quartile Range); unit: MMI (Mean Mass Intensity)
Arm/Group | MEDI4736 + Tremelimumab | Untreated Arm (Control)
Number analyzed (Participants) | 8 | 4
MMI (Mean Mass Intensity) | 0.18 [0.12 to 0.59] | 0.24 [0.11 to 1.08]
Statistical Analysis 1: Comparison: MEDI4736 + Tremelimumab vs Untreated Arm (Control); Compare tumor expression programmed death-ligand 1 (PD-L1) after combination therapy (MEDI-4736 and Tremelimumab) and before and at day 1 of untreated; Test type: Other; p = 0.932, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Median Recurrence-free Survival (RFS)
Description: RFS based on the Kaplan-Meier method is defined as the time between treatment and disease recurrence or censored and participants in either MEDI-4736 alone or MEDI-4736 plus Tremelimumab will be followed up for 2 years after surgery.
Time Frame: Participants will be followed up until disease recurrence or censor for 2 year after surgery
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MEDI4736 | MEDI4736 + Tremelimumab
Number analyzed (Participants) | 8 | 8
months | 14 [3.2 to NA] — The upper 95% confidence limit of the survival curve hasn't reached 50%, there is no estimate for the upper confidence limit on the median. | NA [1.6 to NA] — The median RFS was NA because there was more than 50% survival in the group. The upper 95% confidence limit of the survival curve hasn't reached 50%, there is no estimates for the upper confidence limit on the median.

11. Secondary Outcome: Median Overall Survival (OS)
Description: OS based on the Kaplan-Meier method is defined as the time between treatment and death or censored and participants in either MEDI-4736 alone or MEDI-4736+Tremelimumab will be followed up for 2 years after surgery.
Time Frame: Participants will be followed up until death or censor for 2 year after surgery
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MEDI4736 | MEDI4736 + Tremelimumab
Number analyzed (Participants) | 8 | 8
months | 14.4 [1 to 27] | NA [5.0 to NA] — The median survival was NA because there were more than 50% survival in the group. The upper 95% confidence limit of the survival curve hasn't reached 50%, there is no estimates for the upper confidence limit on the median.

ADVERSE EVENTS:
Time Frame: Adverse events were assessed by the study schedule on the day of infusion and followed up until 4 weeks after hospital discharge, the maximum duration of 24 months
Arm/Group | MEDI4736 | MEDI4736 + Tremelimumab | Untreated Arm (Control)
All-Cause Mortality (participants affected / at risk) | 7/9 | 6/11 | 3/4
Serious Adverse Events (participants affected / at risk) | 4/9 | 4/11 | 1/4
Other Adverse Events (participants affected / at risk) | 6/9 | 7/11 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI4736 (N=9) | MEDI4736 + Tremelimumab (N=11) | Untreated Arm (Control) (N=4)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Death NOS (General disorders) | 3 (3) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden death NOS (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDI4736 (N=9) | MEDI4736 + Tremelimumab (N=11) | Untreated Arm (Control) (N=4)
Anemia (Blood and lymphatic system disorders) | 5 (5) | 3 (3) | 4 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2)
Salivary duct inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 2 (2) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 2 (2) | 2 (2)
Fever (General disorders) | 1 (1) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 2 (2) | 2 (2)
Alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Fibrinogen decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight gain (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight loss (Investigations) | 0 (0) | 0 (0) | 2 (2)
White blood cell decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (6) | 3 (3) | 4 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/51/NCT02592551/Prot_SAP_000.pdf